CLINICAL TRIAL: NCT06487364
Title: Determination of the Minimal Detectable Change and Minimum Clinically Important Change Score of the Parkinson's Disease Questionnaire-8
Brief Title: Determination of the Minimal Detectable Change of the Parkinson's Disease Questionnaire-8
Status: Recruiting | Type: Observational
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Research Assisstant, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Other Study IDs: 2024/78
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Minimal Detectable Change; Minimal Clinically Important Difference; Parkinson Disease Questionnaire-8
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapy Group: There will be only one group in the study. Patients will only be applied to the physiotherapy program recommended by the specialist physician and physiotherapist. It is not possible to apply any additional treatment within the scope of the study.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — A routine physical therapy program prescribed by a specialist physician and physiotherapist will be applied.

SUMMARY:
This study is conducted to determine how many units of improvement the Parkinson's Disease Questionnaire-8 (PDQ-8), used to evaluate the quality of life of Parkinson's patients, should have to express a significant change in the quality of life. Patients for whom a 30-session physiotherapy program is recommended will be included in the study. Patients will be asked to express the change in their quality of life at the end of treatment. The PDQ-8 survey and Global Rating of Patient-Perceived Changes (GRP-PC) forms will be used to determine these changes. Evaluations will be repeated at the beginning of the treatment program and at the end of the 30th session.

ELIGIBILITY:
Inclusion Criteria:

* Having regular neurology follow-up and using medicine;
* Hoehn and Yahr Scale Stage between 1-3 points;
* Mini-Mental State Assessment Score >24 points;

Exclusion Criteria:

* Having a secondary neurological disease;
* Any surgery and/or trauma affecting the upper extremity
* Having complaints of pain before the treatment program;
* There was a change in medical treatment during the study;
* With symptoms of anxiety and depression;
* Those who use alcohol and drugs;
* Individuals with vision defects that cannot be corrected by the use of glasses and those with hearing loss

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson Disease
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
Parkinson Disease Questionnaire-8 | 7 days before the Physiotherapy session
  It is an 8-item form used to assess the quality of life in Parkinson's disease.
Parkinson Disease Questionnaire-8 | First day of the physiotherapy session
  It is an 8-item form used to assess the quality of life in Parkinson's disease.
Parkinson Disease Questionnaire-8 | 6 weeks (5 physiotherapy sessions for 6 weeks)
  It is an 8-item form used to assess the quality of life in Parkinson's disease.

SECONDARY OUTCOMES:
Demographic Data Form | First day of the physiotherapy session
  This form was created by researchers and it consist of personal informations such as gender, education, age, body mass index, duration of disease
Modified Hoehn & Yahr Scale | First day of the physiotherapy session
  It is used to determine the disease stage. It stages the disease between 1 and 5 points. As the stage progresses, disability also increases.
Unified Parkinson's Disease Rating Scale (UPDRS) | First day of the physiotherapy session
  It can assess Parkinson's disease with its different clinical features, including motor and non-motor. It consists of 4 subsections and 55 items in total. This study will use part III of the UPDRS score (between subsections 3.1 and 3.18)
Global Rating of Patient-Perceived Changes (GRP-PC) | 6 weeks (5 physiotherapy sessions for 6 weeks)
  GRP-PC will used to assess patient-perceived hand dexterity changes after the routine intervention. The patient will first asked, "Has your hand dexterity changed compared to when you did not receive interventions?". If the answer is no, the person will given a score of 0 (i.e. no change). In the case of positive response, the patient will asked, "How much better or worse is your hand dexterity" and the patient response will scored on the following 14-point Likert scale: +7 (very much better), +6 (much better), +5 (better), +4 (relatively better), +3 (somewhat better), +2 (a little better), +1 (very little better), -1 (very little worse), -2 (a little worse), -3 (somewhat worse), -4 (relatively worse), -5 (worse), -6 (much worse), and -7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Murat Emirzeoğlu, PhD, Study Chair — Karadeniz Technical University; Adem Aktürk, PhD, Study Chair — İstanbul Gelişim University; Tuğba Eyigürbüz, PhD, Study Chair — Bağcılar Education and Research Hospital
Locations (1):
- Private Güney Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided